CLINICAL TRIAL: NCT05805566
Title: Post-Covid Syndrome Cohort
Brief Title: Retrospective and Prospective Cohort of Patients Entering the Multidisciplinary Management of Post-Covid Syndromes
Acronym: SyPoCo
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_1053
Record Dates: First submitted 2023-04-07; First posted 2023-04-10 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Post-Covid Syndrome
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-Covid Syndrome Patients
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: Blood collection — Blood samples will be collected from the patient at baseline. This blood will be collected during the standard of care blood drawing in extra.

SUMMARY:
SARS-CoV2 pneumonia has been a global public health emergency since 2020. The prevalence of the disease is particularly high with more than 500 million cases worldwide (7.5 million in France) since the emergence of the virus.

A substantial proportion of patients with SARS-Cov2 infection present persistent symptoms long after the acute infection. This is independent of the degree of severity of the SARS-Cov2 infection.

These symptoms can affect the quality of life and impede the return to work. While the majority of symptoms progress favourably with outpatient care, some persist and/or are particularly severe, justifying expert and multidisciplinary care.

This investigation aim to create a clinical database of patients with complex and/or severe post-CoviD and study blood markers what could predict the disease and orientate new ways of treatment.

ELIGIBILITY:
Inclusion Criteria:

All patients who have joined the Epsilon care pathway since its opening in February 2022, i.e.:

* Patients with post-Covid syndrome referred to the Epsilon sector from the city medicine:
* Patient with documented SARS-Cov2 pneumonia
* With persistent and severe symptoms beyond 4 weeks or complex or disabling symptoms beyond 3 months
* Patient over 18 years old.

Post-hospital sector:

* Patient with documented SARS-Cov2 pneumonia
* Hospitalized for oxygen therapy (at least 48h)
* Not having a referring pulmonologist
* Not institutionalized
* With a life expectancy of more than 6 months.

Exclusion Criteria:

* Patient refusing that this data to be used for research purposes (objection form).
* Patient with untreated comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will focus on adult patients with SARS COV2 whose symptoms persist beyond 4 weeks after the acute phase and who will have integrated the Epsilon care system in the pneumology department of Lyon Sud Hospital.
  It is difficult to define an exact number of subjects because this syndrome is still poorly characterized.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Create a patient cohort | Once a year
  Creation of a retrospective and prospective cohort combining:
  * Collection of clinical and paraclinical data, scores, and scales.
  * Prospective monitoring of quality of life, other scores as needed. Cross-referencing of clinical data with the results of cellular and molecular analyzes on lymphocytes blood cells, which will be carried out (part carried out by Inserm). by INSERM U1111 as part of the European HERVCOV project.

SECONDARY OUTCOMES:
Identify new research pathway to improve Post-Covid syndrome knowledge | 12 month
  Description of biological data and clinical and paraclinical data to determine the duration of the syndrome, refine the diagnosis and optimize future management.
Biological analyses to find new molecular targets (biomarkers) | 12 month
  Biological analyzes of blood constituents for the detection of molecular and/or cellular modifications, which could be at the origin of the symptoms (Carried out by Inserm).

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien COURAUD, Pr, Principal Investigator — Department of Acute Pneumology and Thoracic Oncology, Hôpital Lyon Sud, Hospices Civils de Lyon
Locations (1):
- Department of Acute Pneumology and Thoracic Oncology, Hôpital Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite, France